CLINICAL TRIAL: NCT06539247
Title: Comparative Effects of Motor Relearning Approach Versus Proprioceptive Neuromuscular Facilitation Technique (PNF) on Pain, Foot Drop, Gait and Functional Mobility in Hemiplegic Patients
Brief Title: MRP Verses PNF on Pain, Foot Drop, Gait and Functional Mobility in Hemiplegic Patients.
Acronym: CEMRA-PNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Hamna Sarfraz, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec-UOL-/200/08/24
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Pain; Gait, Drop Foot; Foot Drop; Hemiplegia
Keywords: Motor Relearning; Proprioceptive Neuromuscular Facilitation; Muscle Stimulation; Gait Analysis; Functional Mobility
MeSH Terms: conditions — Stroke; Pain; Gait Disorders, Neurologic; Peroneal Neuropathies; Hemiplegia | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Group A: Motor Relearning Approach with EMS Group B: Proprioceptive Neuromuscular Facilitation Technique with EMS
Who Masked: Outcomes Assessor
Masking Description: Single-blinded assessor was considered to minimize bias in outcome measurements. The assessor was unaware of the intervention group assignment for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motor Relearning Approach with EMS (MRA + EMS) (Experimental): This arm received a 30-minute motor relearning program focused on improving foot drop and gait patterns. The program consisted of:
  Motor Relearning Practice (20 minutes): Participants practiced walking, starting with individual components and gradually progressing to full walking sequences. The unaffected leg initiates each step, with the physiotherapist providing support as needed (Singh, 2017).
  Electrical Muscle Stimulation (EMS) for Targeted Activation (10 minutes): EMS applied to the affected ankle dorsiflexors for 10 minutes to stimulate muscle activation. The parameters were:
  Pulse amplitude: 40 mA (default) Pulse duration: adjusted to achieve balanced maximum ankle dorsiflexion Mode: adaptive, considering both intensity and duration for safe foot lift during walking Electrode placement: on the affected ankle dorsiflexors Intensity: set to a comfortable level for the participant (Knutson & Chae, 2010)
  Interventions: Combination Product: Motor Relearning Program with Electrical Muscle Stimulation (MRA + EMS)
- Proprioceptive Neuromuscular Facilitation with EMS (PNF + EMS) (Experimental): This arm received a 30-minute intervention combining Proprioceptive Neuromuscular Facilitation (PNF) techniques and EMS. The program consisted of:
  PNF Techniques for Neuromuscular Facilitation (20 minutes) in side-lying position with the affected leg uppermost. The sequence involved rhythmic initiation movements, measured using an alarm clock (Singh, 2017).
  Electrical Muscle Stimulation (EMS) for Muscle Response Enhancement (10 minutes): Similar to Arm 1, EMS applied to the affected ankle dorsiflexors for 10 minutes with the same parameters:
  Pulse amplitude: 40 mA (default) Pulse duration: adjusted to achieve balanced maximum ankle dorsiflexion Mode: adaptive, considering both intensity and duration for safe foot lift during walking Electrode placement: on the affected ankle dorsiflexors Intensity: set to a comfortable level for the participant (Knutson & Chae, 2010)
  Interventions: Combination Product: Proprioceptive Neuromuscular Facilitation Technique with Electrical Muscle Stimulation (PNF + EMS)

INTERVENTIONS:
Combination Product: Motor Relearning Program with Electrical Muscle Stimulation (MRA + EMS) — This arm received a 30-minute motor relearning program focused on improving foot drop and gait patterns and Electrical Muscle Stimulation (EMS) for Targeted Activation (10 minutes) with 40 mA (default) adaptive, considering both intensity and duration for safe foot lift during walking.
  Arms: Motor Relearning Approach with EMS (MRA + EMS)
Combination Product: Proprioceptive Neuromuscular Facilitation Technique with Electrical Muscle Stimulation (PNF + EMS) — This arm received a 30-minute intervention combining Proprioceptive Neuromuscular Facilitation (PNF) techniques and EMS. The program consisted of:
  PNF Techniques for Neuromuscular Facilitation (20 minutes) and Electrical Muscle Stimulation (EMS) for Muscle Response Enhancement (10 minutes): Similar to Arm 1, EMS applied to the affected ankle dorsiflexors for 10 minutes with the same parameters.
  Arms: Proprioceptive Neuromuscular Facilitation with EMS (PNF + EMS)

SUMMARY:
This single blinded randomized control study aimed to determine the comparative effectiveness of two rehabilitation approaches for improving pain, foot drop, gait, and functional mobility in patients with hemiplegia. The study recruited 68 patients diagnosed with hemiplegia who met specific inclusion criteria. Both groups received a treatment program lasting eight weeks, with assessments at baseline, week four, and week eight. The study measured various outcomes as gait analysis, foot drop grading, functional ability and pain assessment. This study aimed to contribute to evidence-based practice in stroke rehabilitation by comparing the effectiveness of motor relearning and PNF approaches for improving gait, pain, and functional mobility in hemiplegic patients. The findings may help guide therapists in selecting the most appropriate intervention for individual patients.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability worldwide, with hemiplegia (muscle weakness or paralysis on one side of the body) being a common consequence. Rehabilitation plays a crucial role in improving gait, reducing pain and enhancing functional mobility for stroke patients. This study investigated the comparative effects of two rehabilitation approaches: Motor Relearning (MRP) and Proprioceptive Neuromuscular Facilitation (PNF).

Study Design: This was a randomized controlled trial with two parallel groups:

Group A: Motor Relearning Approach with Electrical Muscle Stimulation (EMS) Group B: Proprioceptive Neuromuscular Facilitation Technique (PNF) with Electrical Muscle Stimulation (EMS)

Randomization: Eligible participants were randomly assigned to either group using a lottery method to ensure balance between groups.

Blinding: The assessor evaluating outcomes were blinded to group allocation (single-blinded).

Intervention: Both groups received an eight-week intervention program with assessments at baseline, week four, and week eight. Each session lasted approximately 30 minutes.

Group A (MRP with EMS): Participants performed motor relearning exercises targeting foot drop and gait patterns. EMS was integrated during specific exercises for targeted muscle activation.

Group B (PNF with EMS): Participants received PNF techniques designed to improve neuromuscular facilitation for gait and foot clearance. EMS was used alongside PNF exercises to enhance muscle response.

Outcome Measuring Tools:

Primary Outcomes: Dynamic Gait Index (DGI) for gait analysis and Manual Muscle Testing (MMT) test for foot drop grading Secondary Outcomes: Motor Assessment Scale to measure of functional ability and Numeric Pain Rating Scale (NPRS) for pain assessment.

Ethical Considerations: This study has received ethical approval from the Institutional Review Board (IRB). Informed consent was obtained from all participants.

Data Analysis: Statistical software was used to analyze the data, with appropriate tests employed based on data normality to compare outcomes between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients having age between 45 to 65 years (Kagawa et al., 2013)
* Hemiplegic, impaired functional mobility and dependent (Kanase, 2020)
* Functional deficits in lower limb, with both the Sexes and any side (left or right) (Kanase, 2020)
* Patients having hemiplegia within 6 months might be post-stroke, able to follow instructions (Kanase, 2020)
* Diagnosed with hemiplegia having a stable neurological condition (e.g., stroke) (Anandan et al., 2020)
* Minimum score of 12 on the Dynamic Gait Index (DGI) to ensure sufficient baseline gait function for meaningful comparison (Singha, 2017).
* Grade 3 foot drop (Tibialis Anterior) on the Motor Assessment Scale in the affected leg to have room for improvement in both interventions (Singha, 2017).
* Participants having moderate to severe pain of ≤ 4 (moderate) and ≥ 7 (severe) on numeric pain rating scale (NPRS) at rest , were included to minimize confounding effects of pain on gait and mobility (Beebe et al., 2021).
* Mini-Mental State Examination (MMSE) score ≥ 24 (Page et al., 2007).

Exclusion Criteria:

* Subjects having any medical condition that affects his/her performance (Kanase, 2020)
* Completely recovered case of Hemiplegia in terms of walking abilities & upper limb activities (Kanase, 2020)
* Subjects with Transient Ischemic Attack (Kanase, 2020)
* Other neurological conditions such as severe cognitive impairments

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-01-28 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Gait analysis | 8 weeks (baseline, fourth week and then at the end of the 8 week)
  The Dynamic Gait Index was a standardized tool used to assess gait function in individuals with lower extremity impairments. It evaluated 8 components of gait, with higher scores indicating better gait quality. A total score below 19 suggests a higher risk of falls, whereas scores above 22 are associated with safe ambulation
Foot Drop | 8 weeks (baseline, fourth week and then at the end of the 8 week)
  Manual Muscle Testing was a standardized test that assessed muscle strength on a 5-point scale (0 = no contraction to 5 = normal strength). This was used specifically for the affected leg's dorsiflexor muscles (Tibialis Anterior).

SECONDARY OUTCOMES:
Functional Ability | 8 weeks (baseline, fourth week and then at the end of the 8 week)
  The Motor Assessment Scale is a clinical tool designed to evaluate functional abilities in stroke patients, focusing on everyday motor functions. The scale ranges from a minimum score of 0 (indicating inability to perform tasks) to a maximum score of 6 (indicating optimal performance across all tasks). Higher scores reflect greater functional independence, making it a valuable assessment for rehabilitation settings.
Pain intensity | 8 weeks (baseline, fourth week and then at the end of the 8 week)
  The Numeric Pain Rating Scale is a widely utilized tool for assessing pain intensity in adults. It operates on an 11-point scale ranging from 0 to 10, where 0 indicates no pain and 10 represents the worst pain imaginable. Higher scores on this scale signify greater pain intensity, making it a straightforward method for patients to communicate their pain levels to healthcare providers.

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Sharif, PHD, Principal Investigator — Associate Professor; Hira Riaz, MSOMPT, Study Director — Assistant Professor
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The data was collected from the Sehat Medical Complex, Hanjarwal and University of Lahore Teaching Hospital, Lahore after taking informed written consent form through the questionnaires. A comparative analysis was conducted between Group A and Group B, evaluating improvements in MMT Grading , Dynamic Gait Index, Numeric Pain Rating Scale (NPRS) and Motor Assessment scale scores. The data was entered and analyzed using SPSS Version 24.

REFERENCES:
- [Background] Beebe JA, Kronman C, Mahmud F, Basch M, Hogan M, Li E, Ploski C, Simons LE. Gait Variability and Relationships With Fear, Avoidance, and Pain in Adolescents With Chronic Pain. Phys Ther. 2021 Apr 4;101(4):pzab012. doi: 10.1093/ptj/pzab012. PMID 33482005
- [Background] Kagawa S, Koyama T, Hosomi M, Takebayashi T, Hanada K, Hashimoto F, Domen K. Effects of constraint-induced movement therapy on spasticity in patients with hemiparesis after stroke. J Stroke Cerebrovasc Dis. 2013 May;22(4):364-70. doi: 10.1016/j.jstrokecerebrovasdis.2011.09.021. Epub 2011 Nov 10. PMID 22078779
- [Background] Knutson JS, Chae J. A novel neuromuscular electrical stimulation treatment for recovery of ankle dorsiflexion in chronic hemiplegia: a case series pilot study. Am J Phys Med Rehabil. 2010 Aug;89(8):672-82. doi: 10.1097/PHM.0b013e3181e29bd7. PMID 20531158
- [Background] Page SJ, Levine P, Leonard A. Mental practice in chronic stroke: results of a randomized, placebo-controlled trial. Stroke. 2007 Apr;38(4):1293-7. doi: 10.1161/01.STR.0000260205.67348.2b. Epub 2007 Mar 1. PMID 17332444
- [Background] Anandan, D., PK, T. N., Arun, B., & Priya, V. (2020). Effect of task specific training with proprioceptive neuromuscular facilitation on stroke survivors. Biomedicine, 40(3), 363-366.
- [Background] Kanase, S. B. (2020). Effect of motor relearning programme and conventional training on functional mobility in post stroke patients. Indian Journal of Public Health Research & Development, 11(5), 496-501.
- [Background] Singha, R. (2017). Motor Relearning Program versus Proprioceptive Neuro-Muscular Facilitation Technique for Improving Basic Mobility in Chronic Stroke Patients-A Comparative Study. Int J Physiother Res, 5(6), 2490-2500.